CLINICAL TRIAL: NCT07055568
Title: A Clinical Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of Allogeneic iNKT Cell Infusion in Subjects With Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang Long, Chief physician of hepatobiliary and pancreatic surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250407033053070
Record Dates: First submitted 2025-06-23; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iNKT (Experimental)
  Interventions: Drug: iNKT

INTERVENTIONS:
Drug: iNKT — iNKT: Intravenous infusion, 0.5×10^8cell-3.0×10^8 cell

SUMMARY:
To evaluate the preliminary safety and tolerability of iNKT cell injection after infusion in each group of subjects, and to determine the maximum tolerated dose (MTD) and/or the recommended dose for extended studies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in clinical research; Fully understand this study and voluntarily sign the informed consent form; Willing to follow and capable of completing all the test procedures;
* 2. Male or female, aged 18 to 75 years old (including the boundary value);
* 3. Patients with locally advanced or metastatic pancreatic cancer confirmed by histology or cytology. Patients with locally advanced or metastatic pancreatic cancer that cannot be surgically resected and have failed standard first - or second-line treatments, or have intolerable toxic and side effects of the existing standard treatments, or are not applicable to standard treatments at the present stage, or refuse standard treatments;
* 4. According to RECIST version 1.1, there is at least one evaluable tumor lesion;
* 5. The toxic reactions caused by previous anti-tumor treatment were relieved to grade 0-1 (according to NCI CTCAE version 5.0) or to an acceptable level of the inclusion/exclusion criteria. Except for other toxicities such as hair loss and vitiligo that researchers consider not to pose a safety risk to the subjects;
* 6. Have sufficient organ functions;
* 7. The physical condition score of the Eastern Cooperative Oncology Group (ECOG) in the United States was 0-1;
* 8. The expected survival period is more than 3 months;
* 9. Premenopausal female subjects had negative blood pregnancy results before the start of the study treatment and were willing to abstain from sex or take medically recognized effective contraceptive measures (such as intrauterine devices, condoms) within 6 months from the signing of the informed consent form until the end of the last infusion;
* 10. Male subjects are willing to abstain from sexual activity or take medically recognized effective contraceptive measures for 6 months from the date of signing the informed consent form until the end of the last infusion, and not donate sperm during this period.

Exclusion Criteria:

* 1. Participate in clinical trials of other drugs within 30 days before the first infusion;
* 2. Within 30 days before the first infusion, there is a history of allogeneic or autologous T cell, NK cell and other cell therapy;
* 3. Allergic to any component of iNKT cell injection;
* 4) The following treatments or drugs were received before the first infusion:The use of systemic corticosteroids or immunosuppressive drugs within 14 days before the start of the study treatment, excluding local, intranasal, intraocular, intra-articular or inhaled corticosteroids, or receiving systemic steroid hormone replacement therapy at a dose equivalent to 10mg/d prednisone, Short-term (≤7 days) use of corticosteroids is permitted for prevention (such as allergy to contrast agents) or treatment of non-autoimmune conditions (such as delay-type hypersensitivity reactions caused by exposure to allergens); The attenuated live vaccine was administered within 30 days before the start of the research treatment;
* 5. Brain metastasis or the presence of spinal cord compression;
* 6. The subject is diagnosed with severe autoimmune diseases that require systemic immunosuppressants (including but not limited to: steroids) for treatment, or immune-mediated symptomatic diseases, including ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE), and autoimmune vasculitis (e.g., Wegener's granulomatosis);
* 7. Within 5 years prior to the first infusion, there have been other active malignant tumors, except for those malignant tumors that can be treated locally and have been cured (such as basal cell or squamous cell carcinoma of the skin, superficial or non-invasive bladder cancer, carcinoma in situ of the cervix, intraductal carcinoma in situ of the breast, papillary thyroid carcinoma);
* 8. Within 6 months before the first infusion, the following situations occur: transient ischemic attack, cerebrovascular accident, myocardial infarction, unstable angina pectoris; Congestive heart failure classified as grade III or IV by the New York Heart Association (NYHA); Left ventricular ejection fraction < 50%; Or severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III atrioventricular block, etc. Or use a cardiac pacemaker; The electrocardiogram results show clinically significant abnormalities, or QTcF≥450ms (if the first examination is abnormal, retests can be conducted at least 5 minutes later, and the comprehensive result/average value can be taken to determine the qualification);
* 9. There is a history of interstitial lung disease requiring hormone therapy in the past, or there is currently interstitial lung disease;
* 10. There is effusion in the thoracic cavity, pericardium and peritoneal cavity;
* 11. Within two weeks before the first infusion, there were active bacterial, viral, fungal infections, etc;
* 12. Within 2 weeks before the first infusion, there were uncontrolled concurrent diseases including but not limited to: uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) or poorly controlled diabetes even with standardized treatment;
* 13. Subjects with esophageal or gastric varices that require immediate intervention, intestinal obstruction, or those who, based on the researcher's opinion or after consultation with gastroenterologists or hepatologists, are considered to have a higher risk of bleeding, have evidence of portal hypertension (including splenomegaly found through imaging examinations), or have a previous history of varicose vein bleeding;
* 14. Suffering from active infections, including positive hepatitis B surface antigen [HBsAg] and HBV-DNA > the lower limit of the research center's detection value, positive hepatitis C antibody [HCV-Ab] and HCV-RNA > the lower limit of the research center's detection value; Human immunodeficiency virus (HIV) infection or known positive antibodies for acquired immunodeficiency syndrome (AIDS) and syphilis;
* 15. Combined with severe mental illness, or having a clear history of neurological or mental disorders (such as epilepsy, dementia, schizophrenia, etc.), or having a known history of alcohol abuse, abuse of psychotropic drugs or drug abuse;
* 16. During the screening period or before the start of the research treatment, a fever of unknown cause >38.0°C occurred (except for the fever caused by the tumor as judged by the researcher);
* 17. There is a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* 18. Women who are pregnant or breastfeeding;
* 19. As judged by the researcher, the underlying condition of the subjects may increase their risk of receiving the studied drug treatment, or cause confusion in the interpretation of the toxic reactions and AE that occur;
* 20. Other circumstances where the researcher deems it inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | After 28 days of infusion
  Safety
Maximum tolerated dose (MTD) | After 28 days of infusion
  tolerability

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | About 2 years
  Adverse events up to 12 months of follow-up visit judged by the investigator to be associated with iNKT cell infusion, such as abnormalities or changes in laboratory examinations, physical examinations, vital signs, etc.
Antitumor efficacy-Objective response rate (ORR) | About 2 years
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%). In the event of PR or CR
Antitumor efficacy-Duration of response (DOR) | About 2 years
  The period from the first evaluation of CR or PR to the first evaluation of PD(Progressive Disease) or death of any cause.
Antitumor efficacy-Disease control rate (DCR) | About 2 years
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%).
Antitumor efficacy-Progression-free survival (PFS) | About 2 years
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first.
Antitumor efficacy-Overall survival (OS) | About 2 years
  The period from the first infusion to any cause of death